CLINICAL TRIAL: NCT00166985
Title: The Role of Functional MRI and Doppler Sonography in Assessing Intratumoral Angiogenesis of Endometrial Cancer Patients
Brief Title: The Role of Functional MRI and Doppler Sonography in Assessing Blood Vessel Formation Within the Tumors of Endometrial Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701182
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2004-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer, MRI, Doppler sonography, angiogenesis
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Adenocarcinoma of the endometrium is the fourth most frequent cancer in women. Surgery is the treatment of choice in patients with noninvasive or locally advanced disease. The surgical technique consists of an exploratory laparotomy, with total hysterectomy, bilateral oophorectomy, peritoneal washing, and, in selected high-risk patients, omental and peritoneal biopsies and lymphadenectomy. Therefore, preoperative clinical and instrumental staging of the local spread of disease, as well as local and distant lymph node involvement, represent a critical step in tailoring the extent and the radicalness of surgery.

The role of angiogenesis in cancer growth and metastasis has been gaining much attention for decades. Recent clinical evidence supports this notion. The gradual increase in angiogenesis intensity with tumor progression in malignant melanoma has been reported. Abulafia et al. reported that increasing angiogenicity could be noted from simple hyperplasia, complex hyperplasia, atypical hyperplasia, and Stage IA endometrial carcinoma to invasive endometrial carcinoma. The investigators' research team has shown that incremental angiogenesis could be demonstrated in the tumorigenesis and the possibility of lymph node metastasis in endometrial malignancy. Besides, other growth factors such as vascular endothelial growth factor (VEGF), transforming growth factor- (TGF-), IL-6 and IL-8 have also been reported to correlate with the angiogenesis and the metastasis of endometrial cancer. It seems that tumor angiogenesis of endometrial cancer could be utilized as an important parameter to assess the disease severity of the endometrial cancer.

So, the investigators would like to propose this proposal to focus on the tumor angiogenesis in endometrial cancer patients. There are several purposes in this study. First, the investigators will evaluate and compare tumor angiogenesis surveyed from functional MRI and power Doppler sonography in endometrial cancer patients who receive surgery. Second, the investigators will evaluate whether tumor angiogenesis could be a marker to predict the disease severity of endometrial cancer. Third, the role of functional magnetic resonance imaging (MRI) in endometrial cancer will be elucidated.

DETAILED DESCRIPTION:
Adenocarcinoma of the endometrium is the fourth most frequent cancer in women. Surgery is the treatment of choice in patients with noninvasive or locally advanced disease. The surgical technique consists of an exploratory laparotomy, with total hysterectomy, bilateral oophorectomy, peritoneal washing, and, in selected high-risk patients, omental and peritoneal biopsies and lymphadenectomy. Therefore, preoperative clinical and instrumental staging of the local spread of disease, as well as local and distant lymph node involvement, represent a critical step in tailoring the extent and the radicalness of surgery.

The role of angiogenesis in cancer growth and metastasis has been gaining much attention for decades. Recent clinical evidence supports this notion. The gradual increase in angiogenesis intensity with tumor progression in malignant melanoma has been reported. Abulafia et al. observed that increasing angiogenicity from simple hyperplasia, complex hyperplasia, atypical hyperplasia, and Stage IA endometrial carcinoma to invasive endometrial carcinoma has been found by histopathologic examination. Several articles have reported that transvaginal color and pulse Doppler ultrasound may be helpful blood in the evaluation of various gynecologic tumors. Besides, our previous studies have also shown that incremental angiogenesis could be demonstrated in the tumorigenesis and the possibility of lymph node metastasis in endometrial malignancy. Other growth factors such as vascular endothelial growth factor (VEGF), TGF-, IL-6, and IL-8 have also been reported to correlate with the angiogenesis and the metastasis of endometrial cancer. It seems that tumor angiogenesis of endometrial cancer could be utilized as an important parameter to assess the disease severity of the endometrial cancer.

Determining microvessel density is regarded as a standard procedure to quantitate tumor angiogenesis. However, microvessel density always has been assessed retrospectively and in vitro. Preoperative prediction of the microvessel density would be of value clinically for evaluating severity and progression of disease.

So, we would like to propose this proposal to focus on the tumor angiogenesis in endometrial cancer patients. Endometrial cancer patients who will receive staging surgery will be enrolled in this study. Functional MRI, and transvaginal sonography will be undergone before the surgery in each patient. The angiogenesis-related growth factors will be evaluated later from the surgical specimens. The clinical pathologic items, various angiogenic parameters obtained from the MRI and sonography, and angiogenesis-related factors will be compared and correlated together. There are several purposes in this study. First, we will evaluate and compare tumor angiogenesis surveyed from functional MRI and power Doppler sonography in endometrial cancer patients who receive surgery. Second, we will evaluate whether tumor angiogenesis could be a marker to predict the disease severity of endometrial cancer. Third, we will elucidate the role of functional MRI in endometrial cancer.

Endometrial cancer patients with histopathologic proof who are arranged to receive staging surgery are eligible. All patients will undergo surgery, including total abdominal hysterectomy, bilateral salpingo-oophorectomy, and pelvic and/or para-aortic lymph node dissection or sampling. Surgical specimens will be evaluated for tumor size, histologic grading, depth of myometrial invasion, and presence of lymphovascular emboli and lymph node metastasis. Stage will be determined using the International Federation of Gynecology and Obstetrics classification. Tumors of histologic types other than adenocarcinoma and adenoacanthoma will be excluded. The carcinomas were classified using a three-grade system: grade 1 carcinomas showed glandular formation in more than 95% of the tumor, grade 2 carcinomas showed a solid growth pattern in 5-50%, and grade 3 carcinomas showed a solid pattern in more than 50%. All of the patients who will be enrolled into this study need to sign the consent form and the study protocol will be under the approval of the Institutional Review Board of the patient's hospital.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer patients with histopathologic proof who are arranged to receive staging surgery.
* All of the patients who will be enrolled into this study need to sign the consent form and the study protocol will be under the approval of the Institutional Review Board of the patient's hospital.

Exclusion Criteria:

* Tumors of histologic types other than adenocarcinoma and adenoacanthoma will be excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-09; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan